CLINICAL TRIAL: NCT01179880
Title: A Phase 1/2 Study of E6005 in Japanese Patients With Atopic Dermatitis
Brief Title: A Study of E6005 in Japanese Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E6005-J081-101
Record Dates: First submitted 2010-08-04; First posted 2010-08-11 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: Dermatitis; Atopic
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — methyl 4-(((3-(6,7-dimethoxy-2-(methylamino)quinazolin-4-yl)phenyl)amino)carbonyl)benzoate

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: E6005
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6005 — Four Steps of Ointment Application: Step 1: 0.01% of E6005; Step 2: 0.03% of E6005; Step 3: 0.1% of E6005; Step 4: 0.2% of E6005.
  Arms: 1
Drug: Placebo — Matching placebo for each step
  Arms: 2

SUMMARY:
The safety and pharmacokinetics of topical application with E6005 ointment compared to vehicle will be evaluated in Japanese male patients with atopic dermatitis. Additionally, the efficacy of topical application with E6005 ointment will be explored in Japanese male patients with atopic dermatitis.

ELIGIBILITY:
Inclusion criteria;

* Japanese adult male patients with a confirmed diagnosis of atopic dermatitis according to "Guidelines for Management of Atopic Dermatitis" by the Japanese Dermatological Association.
* Patients with evaluable typical eczema on the back (posterior trunk).
* Patients whose age is equal to or more than 20 and less than 65 at the time of treatment and who can provide written informed consent.

Exclusion criteria;

* Patients complicated with eye symptoms (e.g., cataract, retinal detachment), Kaposi varicelliform eruption, and molluscum contagiosum or impetigo contagiosa.
* Patients who had or have a severe allergy such as anaphylactic shock, anaphylactic reaction and anaphylactoid reaction or allergy/hypersensitivity to E6005 or any of their excipients.
* Patients who received any concomitant ethical drugs or any phototherapies within 14 days prior to Baseline. Subjects are allowed to use external steroids and tacrolimus ointment 8 or more days before Baseline and bland emollients free of medicinal properties (e.g., white petrolatum) throughout the study period.
* Patients with any infection that required hospitalization or intravenous/oral treatment with antibiotic/antiviral/antifungal drug(s) within 28 days prior to Baseline.
* Patients who had or have any malignancy, lymphoma, leukemia, or lymphoproliferative disorders, which dose not include skin cancers (e.g., squamous cell carcinoma or basal cell cancer) that were completely removed and have not metastasized for 5 years.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax will be calculated | Until Day 13
Pharmacokinetic parameter tmax will be calculated | Until Day 13
Pharmacokinetic parameter AUC(0-t) will be calculated | Until Day 13
Pharmacokinetic parameter t1/2 will be calculated | Until Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Fukuoka, Japan

REFERENCES:
- [Derived] Ohba F, Nomoto M, Hojo S, Akama H. Safety, tolerability and pharmacokinetics of a novel phosphodiesterase inhibitor, E6005 ointment, in healthy volunteers and in patients with atopic dermatitis. J Dermatolog Treat. 2016;27(3):241-6. doi: 10.3109/09546634.2015.1093587. Epub 2015 Nov 18. PMID 26581111